CLINICAL TRIAL: NCT02865941
Title: Target Fortification of Breast Milk: The Effect of Different Schedules for Milk Analysis on the Growth and Development of Preterm Infants.
Brief Title: Target Fortification of Breast Milk: How Often Breast Milk Needs to be Measured?
Acronym: TFO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Christoph Fusch, Professor, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016TFO2
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Postnatal Growth Disorder
Keywords: Target Fortification; Breast milk analysis; Nutrition; Macronutrient intake; Protein accretion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 milk analysis (Experimental): 1. Macronutrient content (for protein, carbohydrate and fat content) will be analyzed five times per week, of native breast milk batches which had been prepared for 24 hours feeding.
  2. Routine fortifier will be added to breast milk batches.
  3. Modular products for individual adjustment of protein and/or carbohydrate and/or fat will be given in order to achieve target macronutrient level.
  Interventions: Dietary Supplement: Fortification with modular protein; Dietary Supplement: Fortification with modular carbohydrate; Dietary Supplement: Fortification with modular fat
- 1 milk analysis (Experimental): 1. Macronutrient content (for protein, carbohydrate and fat content) will be analyzed once per week of native breast milk batches which had been prepared for 24 hours feeding.
  2. Routine fortifier will be added to breast milk batches.
  3. Modular products for individual adjustment of protein and/or carbohydrate and/or fat will be given in order to achieve target macronutrient level.
  Interventions: Dietary Supplement: Fortification with modular protein; Dietary Supplement: Fortification with modular carbohydrate; Dietary Supplement: Fortification with modular fat

INTERVENTIONS:
Dietary Supplement: Fortification with modular protein — Modular product supplementation is based on most recent breast analysis done for the participant.
Dietary Supplement: Fortification with modular carbohydrate — Modular product supplementation is based on most recent breast analysis done for the participant.
Dietary Supplement: Fortification with modular fat — Modular product supplementation is based on most recent breast analysis done for the participant.

SUMMARY:
It has been observed that target fortification on different schedules leads to meal to meal variation. It changes the ratio of protein to energy and the percentage of carbohydrate to non-protein energy which may, affect growth. In the past, the investigators have analyzed the outcomes of breast milk composition when target fortification is done with different analysis schedules. The investigators were able to measure the macronutrient intake for different milk analysis schedules via a theoretical model and show that the more frequent schedules reduce the variation of fortified-breast milk, whereas a reduced schedule leads to a high variation of macronutrients. It was observed that, in all the breast milk samples measured twice per week, infants achieved on average the recommended macronutrients in line with current recommendations. Nonetheless, the model only looks at the macronutrient intake and does not investigates the relationship between macronutrient variation and its effect on growth.

The aim of the current study is to compare a frequent schedule of measurement of macronutrient analysis with a reduced schedule of measurement and to study its affect on growth, protein accretion and metabolic parameter.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age < 30 weeks (maternal dates or early fetal ultrasound);
2. Tolerating an enteral intake of ≥100 mL/kg/d for ≥ 24h;
3. Subject is anticipated to receive the intervention for ≥ 3 consecutive weeks after full enteral feeding (≥150 mL/kg/d) has been achieved;
4. Written informed consent has been obtained from the infant's legal representative.
5. Multiple births: Each infant will be included in the study if he/she meets the study criteria, and siblings will be individually randomized to one or other of the treatment arms.
6. Discussion with Most Responsible Physician (MRP) and the staff in order to discuss any potential transfer during the next 7 days.

Exclusion Criteria:

1. Gastrointestinal malformation, major congenital anomalies and chromosomal abnormalities;
2. Babies with enterostoma or short gut syndrome;
3. Infants fed more than 25% of mean caloric intake for a consecutive week with formula milk;
4. Fluid restriction <140 mL/kg/d for ≥ 3 consecutive days;
5. Sepsis - all infants with gram-negative sepsis will be removed from the study;
6. Necrotizing enterocolitis, defined by feeding intolerance associated with positive x-ray findings (pneumatosis intestinalis - Bell Stage 2; air in the biliary tract or free air in the peritoneum - Bell Stage 3);
7. Renal disease, defined by symptoms (oliguria, anuria, proteinuria, hematuria) associated with an increased blood urea nitrogen >10 mmol/L and creatinine of 130mmol/L
8. Participation in another clinical trial that may provide an alternative nutritional intervention, which might affect the outcomes of this study. outcomes of this study;
9. Probability of transfer to another neonatal intensive care unit or level II nursery outside the McMaster Children's Hospital, as discussed with the most responsible physician (MRP)

Max Age: 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Growth during first three weeks of intervention | first three weeks during intervention before 36 weeks of gestation

SECONDARY OUTCOMES:
Daily Nutrient intake (kcal, lactose, protein, fat) measured with conventional milk analysis | from inclusion at postmenstrual age <30 weeks until 36 weeks of gestation
Weight Gain | from inclusion at postmenstrual age <30 weeks until 36 weeks of gestation or discharge
Oxidative stress by 8-Oxo-2'-deoxyguanosine metabolites in urine | from inclusion at postmenstrual age <30 weeks until discharge
  Measured by mass spectroscopy
Protein synthesis analyzed by nitrogen excretion in urine [µmol/mL] | first three weeks during intervention before 36 weeks of gestation
Feeding intolerance questionaire | from inclusion at postmenstrual age <30 weeks until discharge
  volume of gastric residuals, color of gastric residuals, vomiting, abdominal girth, abdominal distention
Fat mass [g] | from inclusion at postmenstrual age <30 weeks until discharge
  Measured with bioelectrical impedance analysis
Lean mass [g] | from inclusion at postmenstrual age <30 weeks until discharge
  Measured with bioelectrical impedance analysis
Head circumference [cm] | from inclusion at postmenstrual age <30 weeks until discharge
  Measured by tape
Body length [cm] | from inclusion at postmenstrual age <30 weeks until discharge
  Measured by length board

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Fusch, MD, PhD, Principal Investigator — McMaster Children's Hospital
Locations (1):
- Faculty of Health Science, McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rochow N, Fusch G, Choi A, Chessell L, Elliott L, McDonald K, Kuiper E, Purcha M, Turner S, Chan E, Xia MY, Fusch C. Target fortification of breast milk with fat, protein, and carbohydrates for preterm infants. J Pediatr. 2013 Oct;163(4):1001-7. doi: 10.1016/j.jpeds.2013.04.052. Epub 2013 Jun 12. PMID 23769498
- [Background] Choi A, Fusch G, Rochow N, Sheikh N, Fusch C. Establishment of micromethods for macronutrient contents analysis in breast milk. Matern Child Nutr. 2015 Oct;11(4):761-72. doi: 10.1111/mcn.12053. Epub 2013 Jun 18. PMID 23782538
- [Background] Fusch G, Choi A, Rochow N, Fusch C. Quantification of lactose content in human and cow's milk using UPLC-tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Dec 1;879(31):3759-62. doi: 10.1016/j.jchromb.2011.09.053. Epub 2011 Oct 6. PMID 22041090
- [Background] Fusch G, Rochow N, Choi A, Fusch S, Poeschl S, Ubah AO, Lee SY, Raja P, Fusch C. Rapid measurement of macronutrients in breast milk: How reliable are infrared milk analyzers? Clin Nutr. 2015 Jun;34(3):465-76. doi: 10.1016/j.clnu.2014.05.005. Epub 2014 May 17. PMID 24912866
- [Background] Fusch G, Mitra S, Rochow N, Fusch C. Target fortification of breast milk: levels of fat, protein or lactose are not related. Acta Paediatr. 2015 Jan;104(1):38-42. doi: 10.1111/apa.12804. Epub 2014 Oct 2. PMID 25213193
- [Background] Rochow N, Landau-Crangle E, Fusch C. Challenges in breast milk fortification for preterm infants. Curr Opin Clin Nutr Metab Care. 2015 May;18(3):276-84. doi: 10.1097/MCO.0000000000000167. PMID 25807355
- [Background] Rochow N, Fusch G, Zapanta B, Ali A, Barui S, Fusch C. Target fortification of breast milk: how often should milk analysis be done? Nutrients. 2015 Apr 1;7(4):2297-310. doi: 10.3390/nu7042297. PMID 25835073
- [Background] Fusch G, Kwan C, Huang RC, Rochow N, Fusch C. Need of quality control programme when using near-infrared human milk analyzers. Acta Paediatr. 2016 Mar;105(3):324-5. doi: 10.1111/apa.13305. Epub 2016 Jan 19. No abstract available. PMID 26663457
- [Background] Choi A, Fusch G, Rochow N, Fusch C. Target Fortification of Breast Milk: Predicting the Final Osmolality of the Feeds. PLoS One. 2016 Feb 10;11(2):e0148941. doi: 10.1371/journal.pone.0148941. eCollection 2016. PMID 26863130
- [Background] Kotrri G, Fusch G, Kwan C, Choi D, Choi A, Al Kafi N, Rochow N, Fusch C. Validation of Correction Algorithms for Near-IR Analysis of Human Milk in an Independent Sample Set-Effect of Pasteurization. Nutrients. 2016 Feb 26;8(3):119. doi: 10.3390/nu8030119. PMID 26927169